CLINICAL TRIAL: NCT03899025
Title: Diagnostics of Scaphoid Fractures With High-Resolution Peripheral Quantitative Computed Tomography - Pilot Study
Brief Title: Diagnostics of Scaphoid Fractures With HRpQCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VieCuri Medical Centre (Other)
Responsible Party: Principal Investigator, Dr. Heinrich Janzing, Principal investigator, VieCuri Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL62476.068.17 / V_FX_SCAPH
Record Dates: First submitted 2017-12-20; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Scaphoid Fracture; Scafoïd; Fracture
Keywords: HRpQCT; high resolution quantitative peripheral CT; Xtreme CT scan; CT scan; Diagnoses Disease; Fracture healing
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: The study will be composed of two subsequent phases, designed to fit within the standard clinical protocol for patients presenting at the emergency department, suspected of having a scaphoid fracture. Briefly, a patient presenting at the emergency department with a clinically suspected scaphoid fracture (by physical examination) will be subjected to standard radiographs followed by cast immobilization. When a fracture is confirmed, a conventional CT is planned within 10 days to assess fracture classification, for which the standard radiographs are insufficient. When no fracture is seen on the initial radiographs, the patient is reevaluated within 10 days after the trauma and physical examination and a conventional CT are performed.
  Based on the CT, a treatment strategy is decided with regular follow up visits. This clinical workup is in accordance with national and regional treatment protocols, as well as with current literature discussed in sections 1.1 and 1.2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected scaphoid fracture (Other): Patients with a suspected scaphoid fracture
  Interventions: Radiation: CT

INTERVENTIONS:
Radiation: CT — CT = computed tomography of the hand/wrist HRpQCT = high resolution peripheral quantitative CT scan of the hand/wrist
  Other Names: HRpQCT

SUMMARY:
The scaphoid bone is the most common fractured carpal bone. Scaphoid fractures represent 2-6% of all fractures and occur mainly in young, active patients aged 15 to 40. The scaphoid bone has an essential role in functionality of the wrist, acting as a pivot. Correct treatment of a scaphoid fracture depends on accurate and timely diagnosis, and inadequate treatment can result in avascular necrosis (up to 40%), nonunion (5-21%) and early osteoarthritis (up to 32%) that may seriously impair wrist function. In addition, impaired consolidation of scaphoid fractures results in longer immobilization leading to significant functional and psychosocial impairment thus having considerable socio-economic consequences and negative impact on the quality of life.

Current diagnostic pathways can take up to two weeks to diagnose (or exclude) a scaphoid fracture, leading to overtreatment in patients with a suspected scaphoid fracture since only 15 to 30% of suspected scaphoid fractures in the Netherlands annually is found to be an actual fracture.

Thus, there is significant room for improvement in the diagnostic pathway of scaphoid fractures.

DETAILED DESCRIPTION:
Scaphoid fractures

The scaphoid bone is the most frequently occurring fracture of the carpal bones. Scaphoid fractures represent 2-6% of all fractures and 90% of all carpal fractures in the Netherlands. Scaphoid fractures typically occur in young, active patients aged 15 to 40 years old. The exact incidence is unknown, but approximately 21,000 scaphoid fractures are suspected in the Netherlands each year. However, only 15 to 30% represent real fractures. Because a significant amount of fractures (up to 65% immediately after injury) remain radiographically occult with conventional radiographic imaging, there is a trend of overtreatment of suspected scaphoid fractures, which means a lot of wrists are immobilized unnecessary.

A scaphoid fracture has potentially far reaching consequences for the patient, considering the unique nature of this bone in the human body, as it articulates with five surrounding bones in the wrist. Because of this, it has an essential role in functionality of the wrist, acting as a pivot. The treatment of scaphoid fractures is found to be a challenge. Failure can result in avascular necrosis (up to 40%), nonunion (up to 21%) of the fracture and subsequently early osteoarthritis (up to 32%). Displaced fractures of the scaphoid bone can lead to an even higher rate of complications.

The results of surgical treatment are variable13 and surgery is often initiated in a late phase of the treatment. Both complicated fracture healing and surgical treatment in a late phase of the treatment have severe socio-economical consequences.

Diagnosis and follow up of scaphoid fractures

The accurate diagnosis of a scaphoid fracture is the first step of successful treatment of this injury. Delay in treatment has been shown to negatively affect outcome, with adequate treatment of a scaphoid fracture increasing union rates from 55% to 90-100%.

However, this knowledge supports the overtreatment-tendency in patients suspected of having a scaphoid fracture at the emergency department. It is estimated that only 15-30% of these patients actually have a scaphoid fracture, 1,3-5 resulting in a substantial number of patients wearing a cast for a limited period of time when they do not need it.

As studies have shown, the clinical evaluation directly after trauma is not capable of reliably proving or excluding a scaphoid fracture. Current clinical practice in the Netherlands consists of conventional X-ray, followed by CT one week later when the initial radiographs are negative, but repeated clinical examination does not exclude scaphoid injury. Other imaging modalities such as MRI or bone scintigraphy are also being used. CT scan gives more useful information about the anatomy of a possible fracture and is more easily available in the Dutch situation than MRI and bone scintigraphy. Aside from the diagnostic delay it is difficult to objectify fracture healing with x-ray, CT scan, MRI or bone scintigraphy. Therefore, there is room for improvement of the arsenal to accurately and timely diagnose and classify scaphoid fractures and to evaluate scaphoid fracture healing.

High resolution peripheral quantitative computed tomography

The current clinical imaging techniques used in the diagnosis of scaphoid fractures as described above lack the resolving power needed for detailed cortical measurements and visualization of the trabecular morphology, for which a spatial resolution lower than 200 µm is needed. The development of high resolution CT scanners with a spatial resolution of 150 to 95 µm enables these measurements, specifically for the extremities. These so-called high-resolution peripheral quantitative CT (HR-pQCT) scanners are smaller and less expensive than current clinical whole body CT scanners. A specific HR-pQCT scanner to visualize and assess trabecular structure of peripheral bones in a clinical (trial) setting is the XtremeCT platform (Scanco Medical AG, Switserland). The most recent iteration of this scanner, the XtremeCT-2, has a voxel size of 61 µm and a spatial resolution of 95 µm, which enables the direct assessment of bone micro-architectural parameters. In addition, after digitalization of the trabecular structure a so called virtual bone biopsy is available, which enables the estimation of bone strength parameters by micro-finite element analysis (µFEA).

Validation and reproducibility studies of both the HR-pQCT scanner as well as µFEA have been performed, and in the last decade widespread experience has been gathered concerning the use of these techniques in (clinical) research.

ELIGIBILITY:
Phase I - Diagnostic phase

Inclusion criteria

In order to be eligible to participate in Phase I of the study, a subject must meet all of the following criteria:

1. Adults (18 years or older) who visit the emergency department of the VieCuri Medical Center Venlo with a clinically suspected scaphoid fracture due to a trauma (<1 week after trauma).
2. Patients who understand the conditions of the study and are willing and able to comply with the scheduled radiographic evaluations and the prescribed treatment and rehabilitation.
3. Patients who signed the Ethics Committee approved specific informed consent form prior to inclusion.

Exclusion criteria

A potential subject who meets the following criterion will be excluded from participation in this study:

1. Patients, who as judged by the principal investigator, are mentally compromised or are unlikely to be compliant with the follow-up evaluations schedule.
2. Patients with a scaphoid fracture at the ipsilateral side in medical history
3. Pregnancy.

Phase II - Follow-up phase

Inclusion criteria

In order to be eligible to participate in Phase II of the study, a subject must meet all of the following criteria:

1. Patients who completed Phase I of the study and have a radiographically confirmed scaphoid fracture on CT or HR-pQCT.
2. Patients who signed the Ethics Committee approved specific informed consent form prior to inclusion.
3. Conservatively treated scaphoid fractures.

Exclusion criteria

A potential subject who meets the following criterion will be excluded from participation in this study:

1. Patients, who as judged by the principal investigator, are mentally compromised or are unlikely to be compliant with the follow-up evaluations schedule.
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-11-28 (Estimated); Study Completion 2020-04-28 (Estimated)

PRIMARY OUTCOMES:
Scaphoid fracture detected on CT or HRpQCT | within 10 days after presentation at the emergency department
  Scaphoid fracture detected on CT or HRpQCT, fracture on one of both scans is considered as a scaphoid fracture

SECONDARY OUTCOMES:
Fracture healing using bone parameters of the HRpQCT | untill 26weeks after fracture
  Fracture healing using HRpQCT
Early change in bone strength as a predictive value for long term (26weeks) functional outcome | untill 26weeks after fracture
  Estimation of bone strengths by micro-finite element analysis (µFEA)
Early change in trabecular structure parameters measured by HRpQCT as a predictive value for long term functional outcome (26weeks) | untill 26weeks after fracture
  Bone micro-architectural parameters are measured by HR-pQCT
Early change in cortical structure parameters measured by HRpQCT as a predictive value for long term functional outcome (26weeks) | untill 26weeks after fracture
  Bone micro-architectural parameters are measured by HR-pQCT

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Janzing, MD, PhD, Principal Investigator — VieCuri MC
Locations (1):
- VieCuri Medical Centre, Venlo, Limburg, Netherlands